CLINICAL TRIAL: NCT02868866
Title: Faith, Activity, and Nutrition: Dissemination in Underserved Communities
Brief Title: Dissemination and Implementation of Faith, Activity, and Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Sara Wilcox, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00036222
Record Dates: First submitted 2016-07-12; First posted 2016-08-16 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Physical Activity, Healthy Eating
Keywords: physical activity; nutrition; fruits and vegetables; faith-based; churches
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intervention (Experimental): Training of church committee followed by 12 months of technical assistance phone calls.
  Interventions: Behavioral: Immediate Intervention
- Delayed intervention (No Intervention): 20 churches are followed but receive no intervention.

INTERVENTIONS:
Behavioral: Immediate Intervention — Committees from 40 churches will be trained in the Faith, Activity, and Nutrition program by Community Health Advisors. The training focuses on helping churches create healthier church environments for physical activity and healthy eating using Cohen's structural model of health behavior as a guide. Each church committee participates in a full-day training and submits a program plan and budget. Churches receive materials to support implementation of the program. After the full-day training, trained churches receive 12 monthly technical assistance calls to help them implement their program plan. The church coordinator receives 8 calls and the pastor receives 4 calls over the 12 months. In Phase 2, the intervention is open to any church in the SC Conference of the United Methodist Church.
  Other Names: Faith, Activity, and Nutrition
  Arms: Immediate intervention

SUMMARY:
This dissemination and implementation study will examine the impact of the Faith, Activity, and Nutrition (FAN) program on both church practices and member behaviors in both a countywide (randomized trial) and statewide (quasi-experimental) study. Guided by two theoretical frameworks, the specific aims of the applied research project are to: 1) examine the adoption and reach of FAN in churches and organizational factors associated with adoption; 2) characterize implementation fidelity and multilevel factors associated with implementation; 3) describe organizational maintenance of FAN and factors associated with maintenance; and 4) study the effectiveness of FAN.

DETAILED DESCRIPTION:
The USC PRC's applied research project will study the dissemination and implementation of an evidence-based program shown previously to significantly increase physical activity and fruit and vegetable intake in churches in South Carolina (Faith, Activity, and Nutrition; FAN). Guided by two theoretical frameworks, the specific aims of the applied research project are to: 1) examine the adoption and reach of FAN in churches and organizational factors associated with adoption; 2) characterize implementation fidelity and multilevel factors associated with implementation; 3) describe organizational maintenance of FAN and factors associated with maintenance; and 4) study the effectiveness of FAN. In Phase 1, churches in a rural county with a high proportion of African American residents will be randomized to receive training in FAN from a community health advisor (n=40) or to be part of a delayed intervention control group (n=20). In Phase 2, a quasi-experimental study will be done with a large religious denomination in SC (churches are not randomized).

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 churches: church in Fairfield County, SC with at least 20 members who regularly attend worship service
* Phase 2 churches: church in the SC Conference of the United Methodist Church
* Members (phase 1): adult who regularly attends church participating in the study

Exclusion Criteria:

* Members (phase 1): under the age of 18
* Members (phase 1): does not regularly attend church participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1807 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Adoption | 12 months
  (# of eligible churches that are trained / # of eligible churches)*100
Reach | 12 months
  (# of church members in trained churches / # of members of all eligible churches)*100
Implementation fidelity | 12 months
  Composite score consisting of implementation of core elements of the intervention
Maintenance | 24 months
  organization maintenance of the intervention based on leader reports

SECONDARY OUTCOMES:
physical activity | 12 months
  Self-reported proportion of members meeting physical activity recommendations using (only for phase 1 of study)
fruit and vegetable intake | 12 months
  Self-reported cups per day of fruits and vegetables (only for phase 1 of study)
Self-efficacy for physical activity | 12 months
  Self-reported self-efficacy for physical activity (average of scale items) (only for phase 1 of study)
Self-efficacy for fruit and vegetable intake | 12 months
  Self-reported self-efficacy for fruit and vegetable intake (average of scale items) (only for phase 1 of study)

OTHER OUTCOMES:
Church environment | 12 months
  Church environmental factors that impede or promote physical activity and healthy eating, assessed through staff observations (only for phase 1 of study)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Wilcox, PhD, Principal Investigator — University of South Carolina
Locations (3):
- United States (3):
  - Clemson University, Clemson, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - Fairfield Behavioral Health Services, Winnsboro, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilcox S, Day KR, Saunders RP, Jake-Schoffman DE, Kaczynski AT, Stucker J, Dunn CG, Bernhart JA. The Faith, Activity, and Nutrition (FAN) dissemination and implementation study: changes in and maintenance of organizational practices over 24 months in a statewide initiative. Int J Behav Nutr Phys Act. 2022 Mar 2;19(1):23. doi: 10.1186/s12966-022-01253-9. PMID 35236373
- [Derived] Wilcox S, Saunders RP, Jake-Schoffman D, Hutto B. The Faith, Activity, and Nutrition (FAN) Dissemination and Implementation Study: 24-Month Organizational Maintenance in a Countywide Initiative. Front Public Health. 2020 May 14;8:171. doi: 10.3389/fpubh.2020.00171. eCollection 2020. PMID 32528919
- [Derived] Wilcox S, Saunders RP, Kaczynski AT, Forthofer M, Sharpe PA, Goodwin C, Condrasky M, Kennedy VL Sr, Jake-Schoffman DE, Kinnard D, Hutto B. Faith, Activity, and Nutrition Randomized Dissemination and Implementation Study: Countywide Adoption, Reach, and Effectiveness. Am J Prev Med. 2018 Jun;54(6):776-785. doi: 10.1016/j.amepre.2018.02.018. Epub 2018 Apr 12. PMID 29656913